CLINICAL TRIAL: NCT03570502
Title: Incidence of Postoperative Pancreatic Fistula in the Resection of the Left Pancreas With a Radiofrequency Assisted Transection Device (RFAT-Pancreas)
Brief Title: Incidence of POPF in the Resection of the Left Pancreas With RFAT
Acronym: RFATPancreas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Rita Quesada, Clinical Trial Monitor, Hospital del Mar
Other Study IDs: 2017/7697/I
Record Dates: First submitted 2018-05-17; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Pancreas Neoplasm; Pancreas Cancer; Pancreatic Adenocarcinoma; Benign Pancreas Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the impact of the Radiofrequency assisted transection on the rate of postoperative pancreatic fistula (POPF) after performing distal pancreatectomies, central pancreatectomies and pancreatic enucleation

DETAILED DESCRIPTION:
Among the different methods for sealing the remaining pancreas, resection and sealing devices assisted by radiofrequency energy (RF) have been used, both in experimental studies and in clinical trials, in order to try to reduce the POPF rate. One of these devices is the Coolinside®, which is approved for this indication and is currently used in selected cases, at the Hospital del Mar, among other centers.

Although there are several published studies based on similar technology, the existing publications on the use of Coolinside® in the pancreas have been made in rat and pig animal models. In particular, the most recent study published by Dorcaratto et al. compares the Coolinside device vs. the mechanical stapler in porcine model when performing distal pancreatectomies. The results suggest that the Coolinside device was more efficient in the control of the POPF than the stapler with a POPF index of 12% vs. 36%.

Therefore, this study aims to obtain more clinical evidence about the use of Coolinside in pancreatic resections within a clinical context.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign or malignant lesions of the pancreas
* Subjected to distal, central pancreatectomy or enucleations of the left pancreas
* Patients ASA (American Society of Anesthesiologists I-III
* Open or laparoscopic approach.

Exclusion Criteria:

* ASA ≥IV patients
* Patients with limitrophic or neuroendocrine lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with benign and malignant pancreatic tumours.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula according the 2016 update of the International Study Group (ISGPS) | 1 month
  "Grade A postoperative pancreatic fistula" is now redefined and called a "biochemical leak," because it has no clinical importance and is no longer referred to a true pancreatic fistula. Postoperative pancreatic fistula grades B and C are confirmed but defined more strictly. In particular, grade B requires a change in the postoperative management; drains are either left in place >3 weeks or repositioned through endoscopic or percutaneous procedures. Grade C postoperative pancreatic fistula refers to those postoperative pancreatic fistula that require reoperation or lead to single or multiple organ failure and/or mortality attributable to the pancreatic fistula.

SECONDARY OUTCOMES:
Sex | Inclusion of the patient in the study
  Gender or the patient (Male/Female)
Age | Inclusion of the patient in the study
  Age of the patient (expressed in years) at the moment of the intervention
Consistency of the pancreas | Inclusion of the patient in the study
  It can be defined as "normal", "soft" or "fibrotic"
Level of jaundice | At the moment of the intervention and during the first week of postoperative period
  Bilirubin level at the moment of the intervention and during the first week of postoperative period
Type of surgical procedure | Inclusion of the patient in the study
  Enucleation, central pancreatectomy or distal pancreatectomy
Laparoscopic or open surgery | Inclusion of the patient in the study
  Laparoscopic or open surgery
Total bleeding | During the intervention
  Measured during the procedure
Size of the pancreatic duct | CT scan prior to surgery
  Size of the main pancreatic duct expressed in mm, measured on the last CT before the procedure
Type of tumour | Diagnosis
  Serous cystadenoma Acinar cystadenoma Ductal adenocarcinoma Acinar cell carcinoma Cystadenocarcinoma of acinar cells Intraductal papillary mucinous neoplasia associated with invasive carcinoma Mixed carcinoma (ductal-neuroendocrine or acinar-neuroendocrine) Cystic mucinous neoplasia associated with invasive carcinoma Pancreatoblastoma Serous cystadenocarcinoma Pseudopapillary-solid neoplasia
Postoperative follow-up | 1 year
  Months of follow-up since the pancreatic procedure
Type of the postoperative complication | 1 month
  Description of the type of complication
Body Mass Index (BMI) | Prior the surgery and during the PO follow-up (1 and 6 months)
  Measured such as: BMI in kg/m^2
Diabetes | Before the precedure and during the PO follow-up (1 and 6 months)
  Does the patient has diabetes before or after the precedure?

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Background] Burdio F, Dorcaratto D, Hernandez L, Andaluz A, Moll X, Quesada R, Poves I, Grande L, Caceres M, Berjano E. Radiofrequency-induced heating versus mechanical stapler for pancreatic stump closure: in vivo comparative study. Int J Hyperthermia. 2016 May;32(3):272-80. doi: 10.3109/02656736.2015.1136845. Epub 2016 Jan 29. PMID 26821683
- [Background] Malleo G, Vollmer CM Jr. Postpancreatectomy Complications and Management. Surg Clin North Am. 2016 Dec;96(6):1313-1336. doi: 10.1016/j.suc.2016.07.013. PMID 27865280
- [Background] Ecker BL, McMillan MT, Allegrini V, Bassi C, Beane JD, Beckman RM, Behrman SW, Dickson EJ, Callery MP, Christein JD, Drebin JA, Hollis RH, House MG, Jamieson NB, Javed AA, Kent TS, Kluger MD, Kowalsky SJ, Maggino L, Malleo G, Valero V 3rd, Velu LKP, Watkins AA, Wolfgang CL, Zureikat AH, Vollmer CM Jr. Risk Factors and Mitigation Strategies for Pancreatic Fistula After Distal Pancreatectomy: Analysis of 2026 Resections From the International, Multi-institutional Distal Pancreatectomy Study Group. Ann Surg. 2019 Jan;269(1):143-149. doi: 10.1097/SLA.0000000000002491. PMID 28857813
- [Background] Lin JW, Cameron JL, Yeo CJ, Riall TS, Lillemoe KD. Risk factors and outcomes in postpancreaticoduodenectomy pancreaticocutaneous fistula. J Gastrointest Surg. 2004 Dec;8(8):951-9. doi: 10.1016/j.gassur.2004.09.044. PMID 15585382
- [Background] Yang YM, Tian XD, Zhuang Y, Wang WM, Wan YL, Huang YT. Risk factors of pancreatic leakage after pancreaticoduodenectomy. World J Gastroenterol. 2005 Apr 28;11(16):2456-61. doi: 10.3748/wjg.v11.i16.2456. PMID 15832417
- [Background] Quesada R, Burdio F, Iglesias M, Dorcaratto D, Caceres M, Andaluz A, Poves I, Castiella T, Sanchez P, Berjano E, Grande L. Radiofrequency pancreatic ablation and section of the main pancreatic duct does not lead to necrotizing pancreatitis. Pancreas. 2014 Aug;43(6):931-7. doi: 10.1097/MPA.0000000000000156. PMID 24977335
- [Background] Dorcaratto D, Burdio F, Fondevila D, Andaluz A, Quesada R, Poves I, Caceres M, Mayol X, Berjano E, Grande L. Radiofrequency is a secure and effective method for pancreatic transection in laparoscopic distal pancreatectomy: results of a randomized, controlled trial in an experimental model. Surg Endosc. 2013 Oct;27(10):3710-9. doi: 10.1007/s00464-013-2952-1. Epub 2013 Apr 13. PMID 23584822
- [Background] Quesada R, Andaluz A, Caceres M, Moll X, Iglesias M, Dorcaratto D, Poves I, Berjano E, Grande L, Burdio F. Long-term evolution of acinar-to-ductal metaplasia and beta-cell mass after radiofrequency-assisted transection of the pancreas in a controlled large animal model. Pancreatology. 2016 Jan-Feb;16(1):38-43. doi: 10.1016/j.pan.2015.10.014. Epub 2015 Nov 18. PMID 26639388
- [Background] Diener MK, Seiler CM, Rossion I, Kleeff J, Glanemann M, Butturini G, Tomazic A, Bruns CJ, Busch OR, Farkas S, Belyaev O, Neoptolemos JP, Halloran C, Keck T, Niedergethmann M, Gellert K, Witzigmann H, Kollmar O, Langer P, Steger U, Neudecker J, Berrevoet F, Ganzera S, Heiss MM, Luntz SP, Bruckner T, Kieser M, Buchler MW. Efficacy of stapler versus hand-sewn closure after distal pancreatectomy (DISPACT): a randomised, controlled multicentre trial. Lancet. 2011 Apr 30;377(9776):1514-22. doi: 10.1016/S0140-6736(11)60237-7. PMID 21529927
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257